CLINICAL TRIAL: NCT05741138
Title: Effect of Routine Physical Therapy With and Without Core Stability Exercises in Patients With Lumbar Radiculopathy. A Randomized Controlled Trial
Brief Title: Effect of Routine Physical Therapy With and Without Core Stability Exercises in Patients With Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hassanjavaid19
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Lumbar Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core strengthening group (Experimental): Group A were given the Standard Physical Therapy Treatment along with core strengthening exercises Core strengthening exercises were carried out in their respective standard positions (were modified according to patient's comfortability)
  Interventions: Other: Core strengthening
- Conventional treatment group (Sham Comparator): Group B were given only Standard Physical Therapy treatment.
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Core strengthening — Plank 1-3 sets of 10-15 reps per side at a slow tempo Side plank Draw in and lift, holding for 5 seconds with purposeful engagement of the core and leg musculature. Keep the head, shoulders, hips, knees and feet in a straight line.
  Bridges - Lie supine with your knees bent and the feet flat on the floor. Lift your pelvis off the ground while supporting on your feet and shoulders. The bridge can be progressed by lifting one foot off the ground end extending the knee Leg rises - Lie on your back with your legs straight and your arms by your sides. Then lift one leg 4 inches of the ground. Your back has to stay flat on the floor. Don't allow it to arch. Alternate. The exercise can be progressed by lifting both legs at the same time.
  Arms: Core strengthening group
Other: Conventional treatment — Hot pack and TENS for 10 minutes (lumbar region and calf muscles) Ultrasound for 10 mins (lumbar region and calf muscles) Gentle passive stretching (calf muscles) Isometric exercises (lumbar region)
  Arms: Conventional treatment group

SUMMARY:
The goal of this Randomized controlled trial was to examine the effect of routine physical therapy with and without core stability exercises in patients with lumbar radiculopathy. The main question it aims to answer is:

• To examine the effect of routine physical therapy with and without core stability exercises in patients with lumbar radiculopathy Participants after reading and signing the consent form were included in study according to eligibility criteria and were allocated in to 2 groups, the Standard Physical Therapy treatment along with core strengthening exercises. Core strengthening exercises were carried out in their respective standard positions (were modified according to patient's comfortability). We measured outcome through different outcome measure tools.

DETAILED DESCRIPTION:
Lumbar radiculopathy (LR) is defined as spinal nerve-related symptoms such as back and leg pain, with variable presence of paraesthesias, reflex changes, and secondary interference of normal activities. Lumbar radiculopathy (LR) is a common debilitating condition of lumbar origin which influences both the general population and athletes alike. Its prevalence has been estimated to be 3-5% of the population, affecting both men and women. Core strengthening exercises (CSE) are used to train, strengthen and condition the core muscles surrounding the middle of the body i.e. the abdomen, hips, pelvis and lower back. CSE trains muscle activity patterns without unnecessarily overloading the tissue, and can help to stabilize the spine. Core strengthening exercises were applied on patient with lumbar radiculopathy and calf pain to see whether it helps to reduce pain or not.

Participants were given consent form and after subjects read and sign the informed consent, they were included in study according to eligibility criteria. 2 groups were included in study, the Standard Physical Therapy treatment along with core strengthening exercises. Core strengthening exercises were carried out in their respective standard positions (were modified according to patient's comfortability). We measured outcome through different outcome measure tools.

ELIGIBILITY:
Inclusion Criteria:

* 45-65 years

Both genders

* Low back pain radiating towards calf for more than 2 months (diagnosed by the orthopedic surgeon)

Exclusion Criteria:

* Patients with Inflammatory, infectious, malign or metabolic diseases
* Patients with osteoporosis, neurological defects, calf muscle hypertrophy, cardiovascular disorders any spinal or leg operations
* Pregnancy

Any traumatic History

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-02-04 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-08-16 (Actual)

PRIMARY OUTCOMES:
Lower extremity functional pain scale (change is being assessed) | Change from baseline after 12 weeks
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals.
Oswestry disability index(change is being assessed) | Change from baseline after 12 weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools
visual analog scale (change is being assessed) | Change from baseline after 12 weeks
  A Visual Analogue Scale (VAS) is one of the pain rating scales. It measures pain at line of 10cm.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Javaid, Principal Investigator — University of Lahore
Locations (1):
- Sehat medical Complex, Lahore, Punjab Province, Pakistan